CLINICAL TRIAL: NCT06667804
Title: The Effect of Laughter Yoga on Blood Glucose Level, Disease Perception and Stress Level in Patients With Type 2 Diabetes;Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Blood Glucose Level, Disease Perception and Stress Level in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HAslan; Hakime Aslan (Other: Inonu University)
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; Laughter Yoga; Glucose; Stress
Keywords: Blood Glucose; Nursing; Laughter Yoga; Diabetes Mellitus; Stress
MeSH Terms: conditions — Diabetes Mellitus | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Randomized cotrolled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga group (Experimental): Laughter yoga group
  Interventions: Other: Laughter yoga
- Control group (No Intervention): No intervention was applied to the patients in the control group.

INTERVENTIONS:
Other: Laughter yoga — Laughter yoga was applied to the experimental group for 4 weeks, 2 days a week, for 8 sessions (each session duration is 30-45 minutes on average). - The researcher is certified as an International Leader of Laughter Yoga. As a nursing intervention, patients with T2DM were made to do laughter yoga by the researcher. The laughter yoga program was conducted online (Google meet online) due to the ongoing COVID-19 pandemic at the time of the study. - The sessions were organized as follows: Monday-Thursday 10:00-10:45, Tuesday-Friday 10:00-10:45, Wednesday-Saturday 10:00-10:45. Participants participated in two sessions that were suitable for them within a week. A participant in a group was not allowed to change days in the following weeks.
  Arms: Laughter yoga group

SUMMARY:
Objective:This study was conducted to evaluate the effect of laughter yoga on postprandial blood glucose level, disease perception and perceived stress level in patients with Type 2 diabetes.

Materials and Methods: The research was carried out as a randomized controlled trial. The population of the study consisted of patients who were followed up with the diagnosis of Type 2 diabetes mellitus in a hospital located in western Turkey. The sample consisted of 100 patients (experimental group = 50, control group = 50) determined by power analysis. In the study, simple randomization was performed to assign patients to groups. Patient Introduction Form, The Brief Disease Perception Scale (B-IPQ), Perceived Stress Scale (PSS) and Blood Glucose Level Registration forms were used to collect data from the patients. The patients in the experimental group were made to do 8 sessions of laughter yoga. The experimental group received 8 sessions (each session lasted 30-45 minutes on average) of laughter yoga, 2 days a week for 4 weeks. Patients were asked to measure and record their blood glucose level before breakfast. The yoga session started 30 minutes after breakfast and after the session was completed, they were asked to measure and record their blood glucose levels again at 120 minutes after breakfast. Blood glucose levels of the patients in the control group were measured before and 2 hours after breakfast, 2 days a week.

DETAILED DESCRIPTION:
Non-pharmacological methods, which are now widely used in nursing care, are accepted as a useful approach to reduce pain, stress and anxiety. In this study, the investigators focused on the therapeutic effect of laughter yoga in individuals with diabetes. In the literature, it has been determined that laughter reduces postprandial blood glucose levels, improves the clinical outcomes of disorders such as inflammation, asthma, cancer and heart disease, reduces anxiety and depression, and the reasons for this are the reduction of physiological stress response. In this study, it was thought that laughter yoga would have an effect on blood glucose value, disease perception and perceived stress level in individuals with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2DM for at least 6 months,
* Able to use computer and/or mobile applications,
* At least primary education graduate,
* Using oral antidiabetic drugs,
* No diagnosed psychiatric illness,
* No communication problems,
* Patients who volunteered to participate in the study were included.

Exclusion Criteria:

* - Using Parenteral Insulin,
* The one who doesn't attend all the yoga sessions,
* Patients with physical conditions that prevent them from participating in laughter yoga sessions (respiratory distress, persistent cough, veritgo, severe heart disease, hemeroid, hernia of any kind, severe back pain, urinary incontinence, epilepsy, bleeding tendency, thrombocytopenia and deformity visible on examination),
* Patients taking medication or other nonpharmacological methods to reduce stress,
* Patients who did not want to participate in the study were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Blood glukose level | two days a week for one month
  Fasting blood glucose was measured before breakfast. Postprandial blood glucose was measured 2 hours after breakfast. Laughter yoga sessions were applied to the patients in the experimental group within this two-hour period.

SECONDARY OUTCOMES:
Perception of Illness and Perceived Stress | one month later
  Perception of Illness (The Brief Disease Perception Scale (B-IPQ)) and Perceived Stress (The Perceived Stress Scale (PSS)) level were collected as pre-test data when the study started. One month later, the scales were reapplied and post-test data were collected.
  In the scoring of the Brief Disease Perception Scale (B-IPQ), 7 items are scored on a Likert-type scale between 0-10. A score between 0 and 70 can be obtained from the scale. As the score obtained from the scale increases, the person's threat perception towards the disease increases negatively.
  A score between 0-56 can be obtained from the Perceived Stress Scale (PSS). There is no cut-off point in the scale, and a higher score indicates that the stress perception of the individual is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aslan H, Akturk U. Demographic characteristics, nutritional behaviors, and orthorexic tendencies of women with breast cancer: a case-control study. Eat Weight Disord. 2020 Oct;25(5):1365-1375. doi: 10.1007/s40519-019-00772-y. Epub 2019 Sep 11. PMID 31512190